CLINICAL TRIAL: NCT06910631
Title: Optimisation du Parcours de Soins Des Enfants fébriles Par l'Utilisation de la CRP Capillaire en Soins Primaires : Protocole d'un Essai Multicentrique randomisé
Brief Title: Optimizing the Care Pathway of Febrile Children Via Capillary C-reactive Protein Assay in Primary Care
Acronym: CRP-CAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: RESPIR/2023/CS-01
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Fever
Keywords: C-reactive protein
MeSH Terms: conditions — Fever

STUDY DESIGN:
Intervention Model Description: Cluster randomized step wedge
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capillary CRP (Experimental)
  Interventions: Other: Capillary CRP
- Control (No Intervention): Prior to Capillary CRP condition

INTERVENTIONS:
Other: Capillary CRP — CRP measured semi-quantitatively using ACTIM-CRP device
  Arms: Capillary CRP

SUMMARY:
Fever is the leading reason for outpatient consultations among children aged 2 to 9 years. The main concern in fever is severe bacterial infection, particularly for younger children. History and clinical examination do not always differentiate viral infections from bacterial infection. In 20% of febrile children, no infectious focus is found after examination and additional tests are necessary. The first one is measuring C-reactive protein (CRP). The results are obtained in several hours on an outpatient basis, causing long delays before starting treatment and often requiring telephone calls or further consultations. Emergency room use is constantly increasing, generating growing tensions within healthcare facilities, yet a large number of visits are avoidable. Among children visiting the pediatric emergency room, parents reported being referred by their primary care physician in approximately 20% of cases for children aged 1 to 5 years and in 30% of cases for children under one year old. The use of capillary medical device to measure CRP in primary care could reduce this referral rate and help relieve overcrowding in emergency rooms, as well as unscheduled consultation centers and medical analysis laboratories. This would result in a streamlined care pathway, saving time for both physicians and patients, as well as reducing the cost of care for the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be a member or beneficiary of a health insurance plan
* Children consulting primary health institutes with fever (temperature ≥ 38°C) requiring CRP testing:

  * Fever > 12h in infants aged 3 to 6 months
  * Fever ≥ 5 days in children over 6 months of age
  * Fever >12h regardless of age, and at the time of consultation, the doctor is concerned about the child's general condition, the tolerance of the fever, or doubts about a bacterial focus (e.g. suspicion of pneumopathy, appendicitis, etc.).
* No severity criteria necessitating immediate hospitalization
* No bacterial infection whose diagnosis is exclusively clinical or identified by other means (e.g. purulent AOM, bacterial angina identified by RDT, etc.).
* Child whose parents and child have been informed about the study, and at least one parent has given consent for their child's participation in the study.
* Enrolment of the child according to their capacity of discernment (for children aged 12 and over, enrolment is essential).
* Child affiliated to or benefiting from a health insurance scheme

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or a study with drug or medical device
* Premature infants under one year of age
* Immunosuppression
* Sunstroke
* Chronic infection
* Malignant pathology
* Autoimmune pathology
* Sickle cell disease
* Child with a central catheter

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Referral rates to any facility equipped for emergency laboratory testing between conditions | Day 1
  Referral: Yes/No as reported by the physician
Referral rates to any facility equipped for emergency laboratory testing between conditions | Day 7
  Referral: Yes/No as reported by the parents

SECONDARY OUTCOMES:
Referral rates to medical biology laboratories between conditions | Day 1
  Referral: Yes/No as reported by the physician
Referral rates to medical biology laboratories between conditions | Day 7
  Referral: Yes/No as reported by the parents
Referral rates to emergency departments between conditions | Day 1
  Referral: Yes/No as reported by the physician
Referral rates to emergency departments between conditions | Day 7
  Referral: Yes/No as reported by the parents
Number complementary tests between conditions | Day 1
  Total number of tests as reported by the physician
Number complementary tests between conditions | Day 7
  Total number of tests as reported by the parents
Type of complementary tests between conditions | Day 1
  Qualitative listing of all further tests classified as: biological (CBC, venous CRP, iono/creatininemia, liver function tests, ECBU, others) or imaging (chest X-ray, abdomino-pelvic ultrasound, urinary and renal ultrasound) as reported by the physician
Type of complementary tests between conditions | Day 7
  Qualitative listing of all further tests classified as: biological (CBC, venous CRP, iono/creatininemia, liver function tests, ECBU, others) or imaging (chest X-ray, abdomino-pelvic ultrasound, urinary and renal ultrasound) as reported by the parents
GP satisfaction on care organization | Day 7
  0-10 visual analog scale
The total duration of GP time between conditions | Day 7
  Minutes: measured as consultation time + examination time and time to inform the family
Parent satisfaction with the care pathway | Day 7
  0-10 numeric scale
Rate of antibiotic prescription between conditions | Day 1
  Antibiotic prescription: Yes/No as reported by the physician
Rate of antibiotic prescription between conditions | Day 7
  Antibiotic prescription: Yes/No as reported by the parents
Duration of fever episode between groups | Day 7
  Days counted upon reaching 24 hours without fever
Cost-consequences between groups | Day 7
  euros
Budget impact analysis | Day 7
  euros

CONTACTS AND LOCATIONS:
Overall Officials: Chloé SIKIRDJI, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (16):
- France (16):
  - MSP OLEA, Bezouce
  - MSP Espace Santé Servian, Béziers
  - MSPU Avicenne, Cabestany
  - MSP de Calvisson, Calvisson
  - MSP de Clarensac, Caveirac
  - MMG de Montpellier, Montpellier
  - MSP Montpellier-Cévennes, Montpellier
  - MMG de Narbonne, Narbonne
  - CHU de Nîmes, Nîmes
  - MMG de Nîmes, Nîmes
  - MSP de Pont Saint Esprit, Pont-Saint-Esprit
  - MSPU Pauline Lautaud, Prades-le-Lez
  - MSP Le Prisme, Remoulins
  - MSP Saint-Laurent d'Aigouze, Saint-Laurent-d'Aigouze
  - MSP Sud Minervois, Saint-Marcel-sur-Aude
  - Mspu La Source, Vergèze

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Upon publication
Access Criteria: The IPD will be made available to other researchers upon reasonable request to the corresponding author

REFERENCES:
- [Derived] Griffiths K, Badin M, Bouvet S, Silvente L, Demattei C, Sikirdji C. Optimising the care pathway of febrile children via capillary C-reactive protein assay in primary care: the CRP-CAP cluster randomised stepped-wedge study protocol. BMJ Open. 2026 Feb 4;16(2):e109414. doi: 10.1136/bmjopen-2025-109414. PMID 41638749